CLINICAL TRIAL: NCT02023164
Title: Multicenter Pilot Study to Assess the Feasibility of Conducting Phase III Trial Comparing IV Cetirizine Injection, 10 mg, to IV Diphenhydramine, 50 mg, for The Treatment of Acute Urticaria
Brief Title: Pilot Phase III Clinical Trial of JDP-205 IV Injection for Treatment of Acute Urticaria
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: JDP Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ETTAU-02; CTN-P4-427 (Other: JDP Therapeutics)
Record Dates: First submitted 2013-12-18; First posted 2013-12-30 (Estimated); Results first posted 2024-02-09 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Acute Urticaria
Keywords: urticaria; allergic reaction; cetirizine; JDP-205
MeSH Terms: conditions — Urticaria; Hypersensitivity | interventions — Cetirizine; Diphenhydramine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Test Drug (Experimental): JDP-205 Injection, 10 mg/mL, 1 mL
  Interventions: Drug: JDP-205 Injection
- Control (Active Comparator): Diphenhydramine Injection, 50 mg/mL, 1 mL
  Interventions: Drug: Diphenhydramine

INTERVENTIONS:
Drug: JDP-205 Injection — Cetirizine, 10mg/mL; a single 1.0 mL injection via intravenous (IV) push over a period of ~2 minutes
  Other Names: Cetirizine; Quzyttir
  Arms: Test Drug
Drug: Diphenhydramine — Diphenhydramine Injection, 50 mg/mL; a single 1.0 mL injection via intravenous (IV) push over a period of ~2 minutes
  Other Names: Benadryl; DPH
  Arms: Control

SUMMARY:
This is a multicenter, parallel group, randomized, double-blind pilot Phase III clinical study of JDP-205 (cetirizine) injection, versus diphenhydramine injection, 50 mg/mL (Benadryl or generic equivalent), in approximately 36 patients with acute urticaria requiring treatment in Hospital Emergency Departments, Urgent Care Centers and Allergy Clinics.

DETAILED DESCRIPTION:
Multicenter, parallel group, randomized, double-blind pilot Phase III clinical study of JDP-205 (cetirizine) injection, versus diphenhydramine injection, 50 mg/mL (Benadryl or generic equivalent), in approximately 36 patients with acute urticaria requiring treatment in Hospital Emergency Departments, Urgent Care Centers and Allergy Clinics. This study will be conducted in 33 patient who either present themselves to the hospital emergency department, allergy clinic or urgent care centers with acute urticaria or developed acute urticaria following a allergen challenge at an allergy clinic.

Following informed consent, eligibility will be established, capturing baseline data including vitals, age, medical history, and medications taken prior to coming to the clinical study site. Following data collection, study subjects will be randomized in a 1:1 ratio to receive study drug of either cetirizine 10 mg IV or diphenhydramine, 50 mg IV. Baseline data including vital signs, the extent of urticaria and erythema, the severity of pruritus, and the level of sedation will be recorded prior to and at 1 hour and 2 hours post study drug administration, and at the time of "Readiness for Discharge". The actual time at which the investigator determines that the subject is ready for discharge (physically and mentally fit) from the study site will also be recorded. At these same time intervals, subjects will be asked to self-rate (recorded by study staff) severity of their pruritus and level of sedation (recorded by study staff).

Twenty-four hours following discharge from the study site, study staff will call the subject to ask them a few short questions to follow-up on the treatment of their acute urticaria. All adverse and serious adverse events experienced by the subjects following informed consent, and all data captured will be recorded in the source documents and/or case report forms.

ELIGIBILITY:
Patients are eligible to be included in the study only if they meet all of the following criteria:

Inclusion Criteria:

* Male or female patients with a diagnosis of acute urticaria associated with an acute allergic reaction to a known (e.g. food, medication, insect bites) or unknown allergen who need treatment with an injectable antihistamine to alleviate their symptoms;
* 18 years of age or older;
* Be willing and able to give informed consent;
* Patients with a Physician Pruritus Severity Score ≥ 1 (determined by the investigator);
* Patients with an Extent of Urticaria/Erythema Score ≥ 1 (determined by the investigator).

Exclusion Criteria:

* Receipt of an investigational drug or device, within the past 30 days;
* Patients in whom an antihistamine may be contraindicated (e.g. narrow angle glaucoma, symptomatic prostatic hypertrophy);
* Patients who, in the opinion of the investigator, may not tolerate an IV injection of diphenhydramine 50 mg, or cetirizine 10 mg;
* Receipt of any antihistamine (H1 antagonist) within the past 4 hours regardless of the route of administration, e.g. diphenhydramine, cetirizine, loratadine, fexofenadine, levocetirizine, desloratadine;
* Receipt of an H2 antagonist within the past 12 hours;
* Receipt of doxepin within the past 48 hours; doxepin is an antidepressant, but it also has antihistamine properties;
* Receipt of steroids by the oral, IV, IM, or inhalational routes route within the past 48 hours to manage an acute allergic reaction;
* Receipt of epinephrine (EpiPen or any other brand) within the past 1 hour;
* Has known allergy to hydroxyzine, cetirizine or levocetirizine, or diphenhydramine;
* Pregnancy or breastfeeding;
* Patients who require epinephrine immediately to manage their acute allergic symptoms;
* Patients who have an acute reaction to medication they are taking (e.g. antibiotics, ACE inhibitors, NSAIDs) and who cannot stop the medication;
* Patients who, based on their medical history or in the opinion of the investigator, have chronic idiopathic urticaria, hereditary angioedema, urticaria refractory to antihistamines, or dermatological disease that interferes with evaluation of a therapeutic response;
* Urticaria not associated with an acute allergic reaction;
* Any condition that in the view of the investigator makes the subject unsuitable for enrollment in this study;
* History of HIV or other known immunodeficiency;
* Major medical or psychiatric illness, other than acute urticaria, at the time of presentation;
* Inability to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2013-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janine North, B.S., Study Director — TerSera Therapeutics LLC
Locations (6):
- United States (2):
  - University of Cincinnati, Department of Emergency Medicine, Cincinnati, Ohio
  - OSU Hospitals, Department of Emergency Medicine, Columbus, Ohio
- Canada (4):
  - Glengarry Memorial Hospital, Independent Practice, Alexandria, Ontario
  - Ottawa Hospital, Civic Campus, Ottawa, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Del Carpio Independent Practice, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment of patients who either present to Hospital Emergency Departments, allergy clinics or Urgent Care Centers with acute urticaria, or develop acute urticaria following allergen challenge at an Allergy Clinic.
Period: Treatment Period
Arm/Group | Test Drug | Control
Started | 16 | 17
Completed | 16 | 17
Not Completed | 0 | 0
Period: 24-Hour Follow-Up
Arm/Group | Test Drug | Control
Started | 16 | 17
Completed | 16 | 15
Not Completed | 0 | 2
Not completed — Lost to Follow-up | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Test Drug: 10 mg/mL, 1 mL
  JDP-205 Injection
- Control: 50 mg/mL, 1 mL
  Diphenhydramine
- Total: Total of all reporting groups
Arm/Group | Test Drug | Control | Total
Number analyzed (Participants) | 16 | 17 | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 17 | 32
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: Years] | 36 (17) | 39 (14) | 37 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 9 | 15
  Male | 10 | 8 | 18
Region of Enrollment [Number; unit: participants]
  Canada | 9 | 10 | 19
  United States | 7 | 7 | 14

OUTCOME MEASURES:

1. Primary Outcome: Extent of Urticaria/Erythema Score (Physician Assessment)
Description: Extent of Urticaria/Erythema Score (Physician Assessment), capturing extent of urticaria/erythema, using the Body Chart (adopted from Burn Chart).
  Extent of Urticaria/Erythema Score is the average of the 2 scores:
  1. Percentage of body area using the body chart (adopted from burn Chart) 0 = none, 1= mild (,25% body coverage), 2 = moderate (25-50% body coverage, 3 = Severe/intense .50% body coverage
  2. Intensity of redness (adopted from PASI) 0 = none, 1 = mile (light pink) 2= moderate (pink), 3 =severe/intense (red)
Time Frame: Baseline, 1 hour, 2 hour, Discharge (up to 4 hours)
Population: Extent of Urticaria/Erythema (Physician Score) 0 = none, 1= mild (patient expresses itchiness, but tolerable and does not scratch, 2 = moderate definite awareness, bothersome, intermittently scratch affected area, 3 = severe difficult to tolerate, scratch vigorously
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Test Drug | Control
Number analyzed (Participants) | 16 | 17
units on a scale
  Baseline | 1.91 (0.61) | 1.74 (0.89)
  1 Hour | 1.53 (0.74) | 1.12 (1.05)
  2 Hour: number analyzed (Participants) | 9 | 10
  2 Hour | 0.89 (0.60) | 1.35 (1.03)
  Discharge | 1.09 (0.55) | 0.97 (0.94)

2. Primary Outcome: Physician Pruritus Severity Score
Description: Physician Pruritus Severity Score based on patient expression of severity of itchiness.
  0= none
  1 = Mild (patient expresses itchiness but tolerable, and does not scratch 2= moderate definite awareness, bothersome, intermittently scratch affected area 3= severe difficult to tolerate scratch vigorously
Time Frame: Baseline, 1 hour, 2 hour, discharge or up to 4 hours post intervention, whichever came first
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Test Drug | Control
Number analyzed (Participants) | 16 | 17
score on a scale
  Baseline Assessment | 2. [1. to 3.00] | 2.00 [0.00 to 3.00]
  1 hour Assessment | 1.0 [0.0 to 2.0] | 1. [0.0 to 2.]
  2 hour Assessment | 1.0 [0.0 to 2.0] | 1.0 [0.0 to 2.0]
  Discharge Assessment | 1.0 [0.0 to 2.0] | 0.0 [0.0 to 2.0]

3. Primary Outcome: Patient Pruritis Severity Score
Description: Patient Pruritis Severity Score based on severity of itching at time of assessment.
  How severly are your hives itching at the moment? 0 = none
  1= mild minimal awareness easily tolerated 2 = moderate definite awareness quite bothersome 3= severe difficult to tolerate
Time Frame: Baseline, 1 hour, 2 hour, discharge or up to 4 hours post intervention, whichever came first
Population: Patient Pruritis Severity Score Some subjects were discharged prior to the 2-hour assessment, resulting in the reduced N at 2 hours.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Test Drug | Control
Number analyzed (Participants) | 16 | 17
score on a scale
  Baseline | 2.19 (0.66) | 2.24 (1.03)
  1 Hour | 0.56 (0.63) | 0.82 (1.01)
  2 Hour: number analyzed (Participants) | 9 | 10
  2 Hour | 0.56 (0.53) | 0.90 (1.29)
  Discharge | 0.50 (0.52) | 0.59 (1.06)

4. Primary Outcome: Composite Acute Urticaria Score Change From Baseline
Description: A composite acute urticaria score, the sum of Extent of urticaria/erythema score (Physician), Physician pruritis score and Patient pruritis severity score. A composite acute urticaria score which the sum of the above three parameters (i.e. 0-9) was calculated post hoc for each patient at each time point and then their score change from the baseline were compared between the two treatment groups. Higher values indicate a worse outcome.
Time Frame: Baseline, 1 hour, 2 hour, Discharge (an average of 1 day)
Population: 33 subjects (100%) completed the following treatment assessments for 1 hour and Discharge 2 hour assessment: 9 participants in the "Test Drug" Arm/Group and 10 participants in the "Control" Arm/Group). Some subjects were discharged prior to the 2-hour assessment, resulting in the reduced N at 2 hours.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Test Drug | Control
Number analyzed (Participants) | 16 | 17
score on a scale
  1-Hour Assessment | -3.13 (1.41) | -3.26 (2.10)
  2-Hour Assessment: number analyzed (Participants) | 9 | 10
  2-Hour Assessment | -4.28 (1.12) | -3.65 (2.21)
  Discharge Assessment | -3.81 (1.12) | -3.82 (2.28)

5. Secondary Outcome: Sedation Scores and Time to Readiness for Discharge
Description: Time from study drug injection to time to readiness for discharge based on composite sedation score at readiness for discharge consist of Physician Sedation Score and Patient Sedation Score
  Physician Sedation Score
  Score ranged from 0 to 4 (0=min, 4=max)
  0 = None (Patient is completely alert. Does not look tired at all), 1 = Mild (Patient sitting/lying comfortably, and looks tired), 2 = Moderate (Drowsy, with occasional eyes closing), 3 = Severe (Asleep, with eyes closed but responds to minor motor stimulation), 4 = Extremely Severe (Asleep; does not respond to minor motor stimulation)
  Patient Sedation Score
  Score ranged from 0 to 4 (0=min, 4=max)
  0 = None (Not drowsy at all), 1 = Mild (Slightly drowsy), 2 = Moderate (Quite drowsy), 3 = Severe (Extremely drowsy), 4 = Extremely Severe (Asleep, cannot self-rate)
  Higher the sedation score = worse outcome
  A composite sedation score which is the sum of the two parameters.
Time Frame: Assessed at discharge or up to 4 hours post intervention, whichever came first data at discharge reported.
Population: A summary of treatment effectiveness as evaluated by the investigators at time of discharge.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Test Drug | Control
Number analyzed (Participants) | 16 | 17
score on a scale
  Physician sedation score at Readiness for Discharge | 0.19 (0.40) | 0.35 (0.49)
  Patient sedation score at Readiness for Discharge | 0.25 (0.45) | 0.71 (0.69)
  Composite sedation score at Readiness for Discharge | 0.44 (0.81) | 1.06 (0.97)

6. Secondary Outcome: Percentage of Patients Requiring Additional Medication
Description: Percentage of Patients Requiring Additional Medication (Rescue Medication)
Time Frame: Baseline, 1 hour, 2 hour, Discharge (an average of 1 day)
Population: Subjects who required additional medication. Rescue medication defined as epinephrine, bronchodilators, and steroids usage.
Measure: Count of Participants; unit: Participants
Arm/Group | Test Drug | Control
Number analyzed (Participants) | 16 | 17
Participants
  Rescue Required at Discharge ]Reported by HCP | 1 | 2
  Additional Rescue Required 24 Hours After Discharged as Reported by Patient: number analyzed (Participants) | 16 | 15
  Additional Rescue Required 24 Hours After Discharged as Reported by Patient | 10 | 13

7. Secondary Outcome: Sedation Scores and Time to Readiness for Discharge HH:MM
Description: Time from study drug injection to time to readiness for discharge based on Physician and Patient Sedation Scores
  Physician Sedation Score:
  0 = None
  1 = Mild 2 = Moderate 3= Severe 4 = Extremely Severe Patient Sedation Score 0= None
  1- Mild 2 = Moderate 3= Severe 4 = Extremely Severe Higher scores = worse outcome
Time Frame: Assessed at discharge or up to 4 hours post intervention, whichever came first data at discharge reported.
Population: A summary of treatment effectiveness as evaluated by the investigators at time of discharge.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Test Drug | Control
Number analyzed (Participants) | 16 | 17
Hours | 1.65 (0.53) | 2.23 (1.20)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from time of informed consent through the 24-hour follow-up *after discharge (an average of 36 hours)
Arm/Group | Test Drug | Control
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/17
Other Adverse Events (participants affected / at risk) | 14/16 | 12/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test Drug (N=16) | Control (N=17)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 1 (1) — Drowsiness
Rash pruritic (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3) — Red plaques, skin redness, pruritis urticaria, rash,
Burning sensation (General disorders) | 1 (1) | 1 (1) — Burning sensation
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) — Constipation
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) — Urticaria
Pruritis (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) — Pruritis
Headache (Nervous system disorders) | 1 (1) | 0 (0) — Headache
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) — Upset stomach
Sedation (Nervous system disorders) | 0 (0) | 1 (1) — Sedation
Lip swelling (Gastrointestinal disorders) | 1 (1) | 0 (0) — Lip swelling
Peripheral swelling (General disorders) | 1 (1) | 1 (1) — Swollen lips and legs; General disorders and administration site conditions
Injection site pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Burning at IV site
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) — Tachycardia
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Tachypnea
Rash (Skin and subcutaneous tissue disorders) | 4 (4) | 2 (2) — Rash
Chills (General disorders) | 1 (1) | 0 (0) — Rigors; General disorders and administration site conditions
Adverse event NOS (General disorders) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Redness
Eye swelling (Eye disorders) | 1 (1) | 0 (0) — Swollen eyes
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Back pain
Swelling face (General disorders) | 0 (0) | 1 (1) — Swelling on face; General disorders and administration site conditions
Respiration abnormal (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
This was a pilot Phase 3 study, therefore a description of the statistical analyses was not documented in a separate Statistical Analysis Plan, and instead, are described within the content of the protocol and within the CSR.

The adverse event data were collected in a non-systematic fashion, consisting of adverse events documented as observed by the study site staff and captured based on verbal communication (phone call) to the patient during the follow-up period.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No